CLINICAL TRIAL: NCT04665804
Title: Effects of Creatine Supplementation as Compared to Glucosamine/Chondroitin Sulfate Supplementation in Addition to Exercise and Physical Therapy in the Management of Knee Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUI/CTR/2020/12
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Creatine; Glucosamine; Electric Stimulation Therapy; Heating

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group A (Creatine Supplementation) (Experimental)
  Interventions: Dietary Supplement: Creatine Supplementation; Other: Supervised Exercise training; Other: Home Exercise Program; Procedure: Electrotherapy + Heating; Procedure: Joint Mobilization
- Experimental Group B (Glucosamine and Chondroitin sulfate Supplementation) (Experimental)
  Interventions: Dietary Supplement: Glucosamine and Chondroitin sulfate supplementation; Other: Supervised Exercise training; Other: Home Exercise Program; Procedure: Electrotherapy + Heating; Procedure: Joint Mobilization

INTERVENTIONS:
Dietary Supplement: Creatine Supplementation — Creatine Supplementation 20g/day for 1 week followed by 5 g/day for 3 weeks
  Arms: Experimental Group A (Creatine Supplementation)
Dietary Supplement: Glucosamine and Chondroitin sulfate supplementation — Glucosamine 500 mg Chondroitin sulfate sodium 400mg 3/day
  Arms: Experimental Group B (Glucosamine and Chondroitin sulfate Supplementation)
Other: Supervised Exercise training — Lower Extremity Resistance Exercise Training Treadmill walking 5-10 min for warm up Strength training: (80% of 8RM)
  3 times supervised exercise for 4 weeks leg press, leg extension, Sit to stand squat (mini squats) Stationary Cycling (Maximum Resistance as per patient tolerance till failure)
  3 sets 8 reps 10-15 s rep rest interval 1-2 min set rest interval
Other: Home Exercise Program — 2 sets of 10 repetitions/day of
  AROM isolated knee extension and knee flexion Isometric isolated knee extension and knee flexion Isometric terminal knee extension Sit to stand squat Isometric knee terminal extension
Procedure: Electrotherapy + Heating — Interferential Current therapy (2P), in combination with heating pad for 20 minutes
Procedure: Joint Mobilization — Tibio-femoral Anterior Glide Tibio-femoral Posterior Glide Patellofemoral Joint Mobilization

SUMMARY:
Osteoarthritis (OA) is one of the most common joint disorders, affecting not only the joints but also the surrounding muscles, which become weak. Resistance exercise reduces pain and improves function in patients with OA of the knee. Nonsteroidal anti-inflammatory drugs (NSAIDs) are widely used by patients with OA to reduce pain and thereby maintain the ability to perform daily activities. However, there is accumulating evidence for a negative effect of NSAIDs, thus many patients with OA are treated with dietary supplementations such as glucosamine and chondroitin sulfate, and some studies show a beneficial effects on cartilage and pain. However, their effect on OA symptoms and cartilage remains controversial. On the other hand creatine supplementation has also been observed to show promising effects when combined with resistance training exercise in the elderly, but the evidence is limited in terms of knee osteoarthritis. For this reason the purpose of this study is to determine the effects of creatine supplementation as compared to glucosamine/chondroitin sulfate in the management of knee osteoarthritis when combined with resistance training exercise.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70 years
* Knee OA with history not less than three months.
* Radiological evidences of grade III or less on Kellgren classification.
* Knee pain on VNRS no more than 8/10

Exclusion Criteria:

* Neuromuscular conditions that may lead to fatigue such as multiple Sclerosis
* Signs of serious pathology (e.g., malignancy, inflammatory disorder, infection).
* History of trauma or fractures in lower extremity.
* Signs of lumbar radiculopathy or myelopathy.
* History of knee surgery or replacement.
* Patients on intra-articular steroid therapy within two months before the commencement of the study.
* Impaired skin sensation.
* Impaired renal function

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-12-06 (Actual); Study Completion 2020-12-06 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 2 weeks
  Visual Analogue Scale was used to measure pain scoring from 0-10 cm on a horizontal 10cm line. A greater score reflects higher pain intensity.
Visual Analogue Scale | 4 weeks
  Visual Analogue Scale was used to measure pain scoring from 0-10 cm on a horizontal 10cm line. A greater score reflects higher pain intensity.
Knee Injury and Osteoarthritis Outcome Score | 2 weeks
  Knee Injury and Osteoarthritis Outcome Score (KOOS) to measure physical function and quality of life. A greater score on Knee Injury and Osteoarthritis Outcome Score reflects good prognosis and outcome and a lower score shows poor prognosis and outcome. the score for Knee Injury and Osteoarthritis Outcome Score is reported in the form of percentage i.e. 0-100%.
Knee Injury and Osteoarthritis Outcome Score | 4 weeks
  Knee Injury and Osteoarthritis Outcome Score (KOOS) to measure physical function and quality of life. A greater score on Knee Injury and Osteoarthritis Outcome Score reflects good prognosis and outcome and a lower score shows poor prognosis and outcome. the score for Knee Injury and Osteoarthritis Outcome Score is reported in the form of percentage i.e. 0-100%.
Knee Joint Range of Motion | 2 weeks
  Knee Joint Range of Motion will be measured via goniometry. It is a continuous scale and a greater score reflects greater angular movement possible at the knee joint, which is measured in degrees.
Knee Joint Range of Motion | 4 weeks
  Knee Joint Range of Motion will be measured via goniometry. It is a continuous scale and a greater score reflects greater angular movement possible at the knee joint, which is measured in degrees.
Body Composition | 2 weeks
  Body Composition was measured via bioelectrical impedance analysis. A greater Phase angle reflects better cellular integrity and smaller phase angle reflects poorer cellular integrity.
Body Composition | 4 weeks
  Body Composition was measured via bioelectrical impedance analysis. A greater Phase angle reflects better cellular integrity and smaller phase angle reflects poorer cellular integrity.
Fall risk | 2 weeks
  Fall risk will be measured via Biodex balance system, and greater score reflects greater fall risk and poorer outcome.
Fall risk | 4 weeks
  Fall risk will be measured via Biodex balance system, and greater score reflects greater fall risk and poorer outcome.
5 repetition sit to stand test | 2 weeks
  Time will be measured to perform 5 repetitions of sit to stand activity. Lesser time means a better score.
5 repetition sit to stand test | 4 weeks
  Time will be measured to perform 5 repetitions of sit to stand activity. Lesser time means a better score.
Modified sphygmomanometer dynamometry | 2 weeks
  Modified sphygmomanometer dynamometry was used to measure muscle strength. Greater score will reflect greater muscle strength. The unit of Modified sphygmomanometer dynamometry used will be mmHg (millimeter of mercury).
Modified sphygmomanometer dynamometry | 4 weeks
  Modified sphygmomanometer dynamometry was used to measure muscle strength. Greater score will reflect greater muscle strength. The unit of Modified sphygmomanometer dynamometry used will be mmHg (millimeter of mercury).

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University Institute of Rehabilitation Sciences., Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No